CLINICAL TRIAL: NCT05030298
Title: Preoperative Radiosurgery in High Grade Glioma: A Phase I Clinical Trial: The NeoGlioma Study
Brief Title: Preoperative Radiosurgery for the Treatment of High Grade Glioma, NeoGlioma Trial
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MC210710; NCI-2021-08848 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 20-013209 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2021-08-23; First posted 2021-09-01 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Malignant Glioma
MeSH Terms: conditions — Glioma | interventions — Radiotherapy; Radiation; Radiosurgery; Temozolomide; Magnetic Resonance Spectroscopy; Specimen Handling; Biopsy

STUDY DESIGN:
Intervention Model Description: The first four patients will be treated by standard of care and all subsequently enrolled patients will undergo preoperative radiosurgery by dose escalation schedule.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (stereotactic biopsy, radiosurgery, surgery) (Experimental): Patients undergo MRI-guided stereotactic biopsy. Within 14 days of registration, patients undergo either standard of care surgery or radiosurgery in 1 fraction. Within 14 days, patients who underwent radiosurgery then undergo surgery. Within 4-6 weeks, all patients then receive standard of care radiation therapy over 30 fraction and temozolomide daily with or without TTF at the discretion of the treating neuro-oncologist. Additionally, patients undergo MRI and blood sample collection and optional biopsy throughout the study.
  Interventions: Radiation: Radiation Therapy; Radiation: Radiosurgery; Procedure: Stereotactic Biopsy; Drug: Temozolomide; Procedure: Tumor Treating Fields Therapy; Procedure: Magnetic Resonance Imaging; Procedure: Biospecimen Collection; Procedure: Biopsy; Procedure: Therapeutic Conventional Surgery

INTERVENTIONS:
Radiation: Radiation Therapy — Undergo radiation therapy
  Other Names: Cancer Radiotherapy; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
Radiation: Radiosurgery — Undergo radiosurgery
  Other Names: Ablation, Radiosurgical; Radiation Surgery
Procedure: Stereotactic Biopsy — Undergo MRI-guided stereotactic biopsy
Drug: Temozolomide — Drug
  Other Names: CCRG-81045; Gliotem; Imidazo[5,1-d]-1,2,3,5-tetrazine-8-carboxamide, 3, 4-dihydro-3-methyl-4-oxo-; M & B 39831; M and B 39831; Methazolastone; RP-46161; SCH 52365; Temcad; Temizole; Temodal; Temodar; Temomedac; TMZ
Procedure: Tumor Treating Fields Therapy — Undergo TTF
  Other Names: Alternating Electric Field Therapy; TTF; TTFields
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; nuclear magnetic resonance imaging; sMRI; Structural MRI
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Biopsy — Undergo biopsy
  Other Names: BIOPSY_TYPE; Bx
Procedure: Therapeutic Conventional Surgery — Undergo surgery

SUMMARY:
This phase I trial finds out the possible benefits and/or side effects of radiosurgery before surgery (preoperative) in treating patients with high grade glioma. Radiosurgery uses special equipment to position the patient and precisely give a single large dose of radiation to the tumor. This method may kill tumor cells with fewer doses over a shorter period and cause less damage to normal tissue. Giving pre-operative radiosurgery may improve the odds of brain tumor control and reduce treatment-related side effects.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the feasibility, safety and maximum tolerated dose (MTD) of preoperative radiosurgery in the treatment of patients with biopsy-proven high-grade glioma prior to conventional therapy.

SECONDARY OBJECTIVES:

I. Acute clinical toxicity profile using Common Terminology Criteria for Adverse Events (CTCAE) version 5 (defined as within 4 weeks of completion of postoperative radiotherapy.

II. Radiographic tumor control at 12 months following surgery (per Response Assessment in Neuro-Oncology [RANO] criteria).

III. Rate of pseudoprogression at first post radiation scan (RANO criteria). IV. Overall survival at 12 months following surgery.

CORRELATIVE RESEARCH OBJECTIVE:

I. Evaluation of the tumor repair pathways triggered by radiation, tumor vascular changes, tumor microenvironment immune profiling, cell cultures, and the creation of orthotopic xenograft models for future study.

OUTLINE: This is a dose-escalation study.

Patients undergo magnetic resonance imaging (MRI)-guided stereotactic biopsy. Within 14 days of registration, patients undergo either standard of care surgery or radiosurgery in 1 fraction. Within 14 days, patients who underwent radiosurgery then undergo surgery. Within 4-6 weeks, all patients then receive standard of care radiation therapy over 30 fraction and temozolomide daily with or without tumor treating fields (TTF) at the discretion of the treating neuro-oncologist. Additionally, patients undergo MRI and blood sample collection and optional biopsy throughout the study.

After completion of study treatment, patients are followed up every 2-3 months for 12 months and then every 3 months for up to 3 years after registration.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Clear clinical and radiographic evidence of primary high grade glioma (HGG) as judged by the Mayo multidisciplinary neuro-oncology team (World Health Organization [WHO] grade III-IV, including glioblastoma) regardless of IDH and MGMT status
* Patients who underwent a previous biopsy confirming high grade glioma are eligible for enrollment
* Planned neurosurgical resection of tumor
* Judged to not be at risk of significant clinical risk (i.e. herniation) with radiation-induced edema prior to resection
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1, or 2
* Negative pregnancy test done =< 14 days prior to registration, for women of childbearing potential only. Patients over 50 years of age who decline pregnancy testing are still eligible without a pregnancy test.
* Ability to complete questionnaire(s) by themselves or with assistance
* Provide written informed consent
* Willing to receive adjuvant radiotherapy at enrolling institution at the time of registration
* Willing to provide tissue and/or blood samples for correlative research purposes

Exclusion Criteria:

* Any of the following:

  * Pregnant women
  * Nursing women who are unwilling to cease during therapy
  * Men or women of childbearing potential who are unwilling to employ adequate contraception
* Prior history of cranial radiotherapy
* Unwillingness to participate in study
* Investigator discretion that enrollment on the study would pose undo harm or risk to the patient
* Non-MRI compatible implanted medical device
* Use of systemic anti-cancer therapy within the previous 3 months
* Medical contraindication to craniotomy and tumor resection
* Pathologic confirmation of grade I-II glioma, brain metastasis, or other brain tumor

  * Note: Patients with a history of grade I-II glioma are eligible if they have only received surgery as treatment and now there is concern for transformation to grade III-IV tumor
* Primary spinal cord glioma or primary brainstem glioma
* Residual tumor of excessive volume or eloquent location per investigator discretion
* Patients who are unwilling or unable to comply with study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2023-05-23 (Actual); Primary Completion 2027-09-15 (Estimated); Study Completion 2027-09-15 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients experiencing any acute grade 3 or greater unplanned adverse event | Up to 4 weeks postoperative radiotherapy
  Assessed per Common Terminology Criteria for Adverse Events (CTCAE) version (v)5.0. The toxicity rate will be estimated using a binomial estimator and a one-sided 95% confidence interval (CI) of the rate will be computed with normal approximation.
Acute clinical toxicity | Up to 4 weeks postoperative radiotherapy
  Assessed per CTCAE v5.0. The maximum grade for each type of acute adverse events will be recorded for each patient. Data will be summarized as frequencies and relative frequencies by treatment arm. Additionally, the relationship of the adverse event(s) to the study treatment will be taken into consideration. Rates will be compared between arms using chi-squared tests.
Maximum tolerated dose (MTD) of preoperative radiosurgery | Up to 4 weeks postoperative radiotherapy
  After the trial is completed, the MTD will be based on isotonic regression. The dose for which the isotonic estimate of the toxicity rate is closest to the target toxicity rate will be selected as the MTD. If there are ties, the higher dose level will be selected when the isotonic estimate is lower than the target toxicity rate; and the lower dose level will be selected when the isotonic estimate is greater than or equal to the target toxicity rate.

SECONDARY OUTCOMES:
Radiographic tumor control | At 12 months post-surgery
  Assessed per Response Assessment in Neuro-Oncology (RANO) criteria. The cumulative incidence of radiographic tumor recurrence will be estimated using a competing risks method (Gooley et al.). The competing risks will be death.
Rate of pseudoprogression | At first post radiation scan
  Assessed per RANO criteria. Data will be summarized as frequencies and relative frequencies overall and by treatment dose. Additionally, the relationship of the pseudoprogression(s) to the study treatment will be taken into consideration.
Overall survival | At 12 months post-surgery
  Overall survival (OS) is defined as the time from study enrollment to death by any cause. Will be estimated with a Kaplan-Meier estimator and curve for patients treated with preoperative radiosurgery. Estimates will be given for specific time points along with 95% CIs.

OTHER OUTCOMES:
Tumor tissue evaluation of tumor changes | Up to 14 days Post-radiosurgery
  Any excess tissue recovered from the surgical specimen (after standard of care pathologic evaluation) will undergo a series of advanced testing, potentially including but not limited to evaluation of the tumor repair pathways triggered by radiation, tumor vascular changes, tumor microenvironment immune profiling, cell cultures, and the creation of orthotopic xenograft models for future study. Analysis will be completed outside the scope of this protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel M. Trifiletti, MD, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic in Arizona, Phoenix, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials